CLINICAL TRIAL: NCT06268262
Title: Surgical-imaging Combined Research on Obesity
Brief Title: Surgical-imaging Research on Obesity (SIRO)
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2023-KL045-01
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Overweight; MRI; Bariatric surgery; Fatty liver
MeSH Terms: conditions — Overweight; Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples, biopsied liver tissue, biopsied fat tissue, gastric tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: Non-intervention
- Healthy control: Non-intervention

SUMMARY:
The global obesity epidemic is well established, and is an important public health issue. The previous researches had applied the clues that obesity is a kind of systemic disease. The investigators hypothesized that a serious alteration of the body systems will occur after bariatric surgery, which may shed light on the mechanisms of obesity. Thus, the research aims to combine the imaging and surgery to investigate the alterations of the body that induced by obese and alterations after surgery.

DETAILED DESCRIPTION:
In 2016, the prevalence of obesity has already reached 13% of obesity and about 40% overweight worldwide. There is no doubt that obesity is linked to a broad spectrum of diseases，such as cardiovascular diseases, fatty liver diseases, polycystic ovarian syndrome and even central nervous systems disorders. For instance, in a review, author indicated the insulin resistance of T2DM occurs primarily in the muscles of lean individuals before they become obese. The central nervous system, especially the hypothalamus, has always considered to be the regulation center of food intake and hormonal regulation of energy homeostasis. In turn, obesity may worsen the regularity function of nervous system in several pathway. Based on the previous findings, the investigators hypothesized that a serious alterations of the body systems will occur after bariatric surgery, which may shed light on the mechanisms of obesity. The investigators plan to integrate the MR imaging, biological and epidemiological data thoroughly to investigate the alterations of the body that induced by obese and also followup the alterations that after surgery.

ELIGIBILITY:
Inclusion Criteria for obesity group:

Meeting the obesity criteria (BMI > 28); 2) Meeting the indications for bariatric surgery, planning to undergo surgery for the first time; 3) Age between 18-65 years old, no gender restrictions; 4) Right-handed, of Han ethnicity; 5) Informed consent to the study, willing to cooperate with the research, and able to sign an informed consent form.

Inclusion Criteria for the Control Group:

1. Healthy volunteers with a BMI between 18.5-23.9;
2. Age between 18-65 years old, no gender restrictions;
3. Right-handed, of Han ethnicity;
4. Informed consent to the study, willing to cooperate with the research, and able to sign an informed consent form.

Exclusion Criteria for obesity group:

1. Secondary obesity caused by other organic diseases or medication (such as hormone use, etc.);
2. Unable to undergo surgery as planned;
3. Pregnant or breastfeeding;
4. Low cognitive ability and incapable of cooperating with the study;
5. Eating disorders;
6. Alcohol or drug dependence;
7. Meeting the criteria for organic mental disorders, severe mental disorders (schizophrenia, etc.), or other serious mental illnesses requiring clinical intervention;
8. Contraindications for MR scanning (pacemakers, cochlear implants, metal objects in the body, claustrophobia, weight exceeding the machine's load limit, etc.);
9. History of neurological organic diseases (brain tumors, epilepsy, cerebrovascular accidents, severe head trauma, etc.);
10. History of congenital heart disease (myocardial infarction, severe arrhythmias, heart failure, cardiomyopathy, rheumatic heart disease, congenital heart disease, etc.);
11. Severe liver, kidney, lung, digestive dysfunction, endocrine, and blood system diseases;
12. Active infections within the last two weeks (fever, upper respiratory infection, acute gastroenteritis, etc.);
13. Use of drugs affecting the nervous system or psychotropic drugs within the last six months.

Exclusion Criteria for the Control Group:

The same criteria as points 3) to 13) above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aged between 18 and 65, regardless of gender. Initially diagnosed as obesity (BMI>28) and plan to undergo bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Imaging parameters of obesity | baseline, 6th month
  Brain cortical thickness in millimeter
Imaging parameters of obesity | baseline, 6th month
  The volume of left ventricle in cubic millimeter
Imaging parameters of obesity | baseline, 6th month
  Fat fraction of liver (dividing the in-phase fat attenuation signal by the out-phase fat attenuation signal)

SECONDARY OUTCOMES:
Neurotransmitter, inflammatory factors and hormones related to obesity in blood sample | baseline, 6th month
  The level of 5-HT，GABA, TNF-a and estradiol in ng/L
Neurotransmitter, inflammatory factors and hormones relating to obesity in blood sample | baseline, 6th month
  The level of BDNF in ng/ml
Neurotransmitter, inflammatory factors and hormones related to obesity in blood sample | baseline, 6th month
  cortisol in μg/L
Genetic information from venous blood sample, biopsied liver tissue, biopsied fat tissue, and gastric tissue | baseline
  Screen and analyzing the DNA and RNA related to obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tutor AW, Lavie CJ, Kachur S, Milani RV, Ventura HO. Updates on obesity and the obesity paradox in cardiovascular diseases. Prog Cardiovasc Dis. 2023 May-Jun;78:2-10. doi: 10.1016/j.pcad.2022.11.013. Epub 2022 Dec 5. PMID 36481212
- [Background] Malone JI, Hansen BC. Does obesity cause type 2 diabetes mellitus (T2DM)? Or is it the opposite? Pediatr Diabetes. 2019 Feb;20(1):5-9. doi: 10.1111/pedi.12787. Epub 2018 Nov 5. PMID 30311716
- [Background] Schwartz MW, Woods SC, Porte D Jr, Seeley RJ, Baskin DG. Central nervous system control of food intake. Nature. 2000 Apr 6;404(6778):661-71. doi: 10.1038/35007534. PMID 10766253
- [Background] Raji CA, Meysami S, Hashemi S, Garg S, Akbari N, Gouda A, Chodakiewitz YG, Nguyen TD, Niotis K, Merrill DA, Attariwala R. Visceral and Subcutaneous Abdominal Fat Predict Brain Volume Loss at Midlife in 10,001 Individuals. Aging Dis. 2024 Aug 1;15(4):1831-1842. doi: 10.14336/AD.2023.0820. PMID 37728587
- [Background] Gutierrez-Cuevas J, Santos A, Armendariz-Borunda J. Pathophysiological Molecular Mechanisms of Obesity: A Link between MAFLD and NASH with Cardiovascular Diseases. Int J Mol Sci. 2021 Oct 27;22(21):11629. doi: 10.3390/ijms222111629. PMID 34769060